CLINICAL TRIAL: NCT05388630
Title: The Impact of a Gut-derived Metabolite on Anxiety Behavior of Human Subjects Based on Their Cognitive Orientation Variation
Brief Title: Microbiome, Anxiety and Cognitive Orientation Study
Acronym: MACO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Endominance (Industry)
Collaborators: Dr. John J. Ratey (Unknown); HEM Pharma Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 04012022
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Anxiety; Microbiome; Mood Disorders; Neurodegeneration; Depression
Keywords: Lifestyle; Gut bacteria; 4-ethylphenyl sulfate 4EPS; Cognitive Orientation; Gut Brain Axis; Microbiome; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders; Nerve Degeneration; Depression; Orientation, Spatial

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 4-ethylphenyl sulfate (4EPS) is a molecule produced by gut microbes in mice and humans. An enzyme in the colon and liver converts 4EP to 4EPS, allowing it to circulate in the blood. Research has shown that higher 4EPS levels may strongly be associated with anxiety levels in both humans and mice, through its degenerative effects on oligodendrocyte function and myelin patterning in the brain. This metabolite can be measured in stool and blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mounting evidence shows that the gut microbiome plays an important role in communication within the gut-brain axis. However, the relationship between gut microbiota and their influence on anxiety is still not fully understood. Recent studies on mice found a specific microbe-produced molecule, 4-ethylphenyl sulfate (4EPS), can induce anxious behavior. 4EPS is produced by gut microbes in mice and humans. Research suggests higher 4EPS levels may strongly be associated with anxiety levels. However, anxiety is far more complicated than changes in a single molecule. There are many more factors to consider when it comes to anxiety, including various aspects of one's lifestyle and how humans perceive their environment (cognitive orientation). The primary research goal is to better understand the effects 4EPS has on human anxiety behavior and the role cognitive orientation has in connection to anxiety.

DETAILED DESCRIPTION:
This study aims to expand and improve upon previous research on gut bacteria and their connections to anxiety. The Investigators will examine the gut microbiota and its vital role in the gut-brain axis, the link between a gut-derived bacteria (4EPS) and anxiety, and the connections between cognitive orientation and anxiety. It is hypothesized that even though higher 4EPS levels may be associated with anxiety levels in humans, such levels may be more prominent (severe) or less pronounced (less severe) in humans with variations in lifestyle and cognitive orientation.

Cross-sectional data will be compiled from a cognitive assessment (COSEC), a health/lifestyle survey, a generalized anxiety questionnaire, a depression questionnaire, and a stool sample. Stool samples will be analyzed for 4EPS levels. Using the COSEC assessment, we will divide the subjects into nine groups of unique cognitive styles based on their perception and conception scores. Then, depending on their 4EPS level and their survey responses, the relationship between the level of 4EPS and their cognitive traits will be analyzed. COSEC is a cognitive propensity and behavioral preference diagnostic tool designed to understand people's various tendencies that occur during the process of perceiving the environment and responding in action.

The long-term goal of this project is to find connections in the gut-brain axis and gain a deeper understanding of microbiome metabolites as neurodegenerative agents, as they affect anxiety levels in humans. No other studies have been performed to date combining these research areas or their impacts on humans.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age and older
* Participants must be able to read and write English
* Participants must be able to provide consent independently
* Participants must provide a legitimate postal address/P.O Box
* Participants must have access to a device such as a computer or a smartphone

Exclusion Criteria

-Unable to provide a stool sample due to health status or functional impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nationwide population of adults 18 years of age and older. Participation is fully remote.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-04-11 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
4EPS | up to 2 weeks
  Stool samples will be lab processed and analyzed for 4-EPS levels
Cognitive Orientation Social-Emotional Competency (COSEC) Assessment | up to 1 week
  An online cognitive propensity and behavioral preference diagnostic tool. COSEC is designed to understand people's various tendencies that occur during the process between perceiving the environment and responding in action. It illustrates an individual's personality and aptitude as an outcome shaped by their environment and the perception of the world around them.
  COSEC incorporates the environmental impact on the individual by looking at the unique process of a person's perception, conception, and behavior process. Assessments are scored using an algorithm to generate quantified measurements based on multifactorial relationships between a subject's responses. Results are presented in a descriptive format, called the COBI Report (Cognitive Orientation Behavior Inventory).
Anxiety Assessment | up to 1 week
  GAD-7: Generalized Anxiety Disorder 7 is a self-reported questionnaire for screening and severity measuring of generalized anxiety disorder. Scores of 5, 10, and 15 represent cut points for mild, moderate, and severe anxiety, respectively.
Depression Assessment | up to 1 week
  PHQ-9: Patient Health Questionnaire is a self-administered, 9 question diagnostic tool that rates depression using 9 DSM-V criteria for depression based on the mood.A PHQ-9 score total of 0-4 points equals "normal" or minimal depression. Scoring between 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression.
Lifestyle and Health Survey | up to 1 week
  Demographic, health, and lifestyle data.

CONTACTS AND LOCATIONS:
Locations (1):
- Endominance Inc., Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No
All data will be anonymized and shared in aggregate data sets.

REFERENCES:
- See also: Research Study Landing Page — http://www.endominance.com/maco_study/